CLINICAL TRIAL: NCT02175420
Title: Role of BCG Vaccination as Booster on Salmonella Typhi Vaccine
Brief Title: Role of BCG as Booster Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BCG-TFV1
Record Dates: First submitted 2014-06-20; First posted 2014-06-26 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: BCG Vaccination
Keywords: BCG; Salmonella; Trained immunity; Non-specific effect vaccines
MeSH Terms: interventions — BCG Vaccine; Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TFV alone (Active Comparator): Typhim Vi
  Interventions: Biological: TFV
- BCG+TFV (Experimental): BCG (SSI, Denmark) followed after 14 days by Typhim Vi
  Interventions: Biological: BCG; Biological: TFV

INTERVENTIONS:
Biological: BCG
  Other Names: BCG vaccine (SSI, Denmark)
  Arms: BCG+TFV
Biological: TFV
  Other Names: Typhim Vi

SUMMARY:
The BCG (bacillus Calmette-Guerin) vaccine is used for the protection against tuberculosis.

Apart from it's protective effect against tuberculosis BCG vaccine has been shown to have non-specific effects on the innate immune system and is in epidemiological studies associated with reduced mortality due to infectious diseases.

Several studies have shown that BCG can boost the effect of other vaccines. The present study aims to investigate the boosting effect of BCG on the response to typhoid fever vaccine (TFV) and to assess the non-specific effects of BCG on the innate immune system at early timepoints by vaccinating volunteers with either TFV alone or BCG followed by TFV 14 days later.

The study hypothesis is that when BCG is given 14 days before typhoid fever vaccine a better vaccination result in terms of antibody production will be accomplished against typhoid fever due to the effects of BCG on the innate immune system.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Born in Salmonella typhi endemic country
* Pregnancy
* Oral medication except anticonceptive drugs
* Previous vaccination with BCG and/or TFV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
anti-salmonella typhi Vi antigen antibody titer 2 weeks post TFV | 2 weeks
  anti-salmonella typhi Vi antigen antibody titers at 2 weeks after TFV will be compared between TFV only and TFV after BCG groups.
anti-salmonella typhi Vi antigen antibody titer 3 months post TFV | 3 months
  anti-salmonella typhi Vi antigen antibody titers at 3 months after TFV will be compared between TFV only and TFV after BCG groups.

SECONDARY OUTCOMES:
Change in ex vivo cytokine responses | 0, 1 and 4 days; 2 weeks, 3 months
  Ex vivo cytokine response to unrelated antigens

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Netea, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

REFERENCES:
- [Derived] Blok BA, Arts RJW, van Crevel R, Aaby P, Joosten LAB, Benn CS, Netea MG. Differential effects of BCG vaccine on immune responses induced by vi polysaccharide typhoid fever vaccination: an explorative randomized trial. Eur J Clin Microbiol Infect Dis. 2020 Jun;39(6):1177-1184. doi: 10.1007/s10096-020-03813-y. Epub 2020 Feb 17. PMID 32065303